CLINICAL TRIAL: NCT03108222
Title: Phosphorus Absorption in Healthy Adults and in Patients With Moderate Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Kathleen Hill Gallant, Principal Investigator, Purdue University
Other Study IDs: 1612460566
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Kidney Disease Mineral and Bone Disorder
Keywords: chronic kidney disease; CKD; renal failure; phosphorus; phosphate; intestinal absorption
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects: Healthy subjects, free of CKD
  Interventions: Other: Phosphorus Absorption Test
- Moderate CKD Subjects: Subjects with moderate-stage CKD
  Interventions: Other: Phosphorus Absorption Test

INTERVENTIONS:
Other: Phosphorus Absorption Test — Subjects will undergo a radiophosphorus (P-33) absorption test over two days, that will include an oral administration of P-33 on the 1st day of the test, and an IV administration of P-33 on the 2nd day of the test. P-33 activity from serial serum and urine collections will be determined by scintillation counting, and fractional phosphorus absorption calculated by kinetic modeling.

SUMMARY:
Chronic kidney disease (CKD) affects approximately 26 million Americans with many more at risk for disease development. Elevated serum phosphorus (P) and related abnormalities in P homeostasis due to progressive loss of kidney function are primary driving forces behind cardiovascular dysfunction and mortality in CKD patients. Intestinal P absorption is an critical aspect in P homeostasis but has been understudied, particularly in the early stages of CKD progression. This study aims to determine P absorption in patients with moderate CKD compared to healthy adults.

ELIGIBILITY:
Inclusion:

Men and women ages 30-75 years old, any race

Moderate CKD, based on the last set of labs done in the past year, defined as:

Glomerular Filtration Rate (GFR) category G3a (eGFR 45-59 mL/min) with A2 or A3 albuminuria or proteinuria by positive dipstick or urine protein/creatinine ratio (UPCR); -or- G3b (eGFR 30-44 mL/min), with or without evidence of albuminuria (any A1-A3) or proteinuria. (Figure 1)

-or- Healthy control with no diagnosis or evidence of CKD

Female subjects must be post-menopausal, surgically sterile, or confirmed not pregnant by pregnancy test and not breastfeeding.

Subjects must be on stable doses of medications (except those noted in exclusion criteria) for at least 6 weeks prior to the study

Exclusion:

Plans to initiate dialysis within 6 months

Labs based on the last set done in the past year:

Hypercalcemia defined as serum calcium > 10.5 mg/dL

Hyperkalemic > 5.5 mg/dL Prescribed a phosphate binder medication

Small bowel resection, bariatric surgery. Medically unstable or poorly controlled hypertension, diabetes, or gastrointestinal disorders in the opinion of the physicians on the study team

Calcitriol, ergocalciferol, cholecalciferol, vitamin D analogs, calcimimetics, PTH analogues, calcium supplements, multivitamins/mineral and other medications that may alter phosphorus metabolism - must be off for at least 6 weeks prior to study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and subjects with moderate CKD will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Fractional Phosphorus Absorption | Measured from serial blood draws over a 4-hour time frame
  Radiophosphorus (P-33) activity determined by liquid scintillation counting in serum and urine after oral and IV administration will be used to determine fractional phosphate absorption.

SECONDARY OUTCOMES:
Serum FGF23 | Measured from baseline measures and serial blood draws over a 4-hour time frame
  serum intact and c-terminal FGF23
Serum 1,25(OH)2D | Measured from baseline measures and serial blood draws over a 4-hour time frame
  serum 1,25-dihydroxyvitamin D
Serum parathyroid hormone (PTH) | Measured from baseline measures and serial blood draws over a 4-hour time frame
  serum intact parathyroid hormone
Serum phosphate | Measured from baseline measures and serial blood draws over a 4-hour time frame
  serum phosphate
24h Urine phosphate | measured from two, 24-hour urine collections
  24h urine phosphate

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University Nutrition Science Department, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stremke ER, Wiese GN, Moe SM, Wastney ME, Moorthi RN, Hill Gallant KM. Intestinal Phosphorus Absorption in Moderate CKD and Healthy Adults Determined Using a Radioisotopic Tracer. J Am Soc Nephrol. 2021 Aug;32(8):2057-2069. doi: 10.1681/ASN.2020091340. Epub 2021 Jul 8. PMID 34244325